CLINICAL TRIAL: NCT06666491
Title: A Randomized, Open-label, Multi-center, Interventional Phase 3 Study of the Efficacy and. Safety of Tafenoquine Compared to Primaquine (Both Co-administered With Chloroquine) for the Radical Cure (Relapse Prevention) of Plasmodium Vivax (P. Vivax) Malaria in Indian Participants (Pediatric and Adult Population)
Brief Title: An Interventional Study to Compare the Efficacy and Safety of Tafenoquine (TQ) and Primaquine (PQ) When Either Are Taken Together With Chloroquine (CQ) for the Treatment of P. Vivax Malaria in Indian Participants Aged 2 Years and Older
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 208550
Record Dates: First submitted 2024-10-18; First posted 2024-10-30 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Malaria, Vivax
MeSH Terms: conditions — Malaria, Vivax | interventions — tafenoquine; Primaquine; Chloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQ/CQ (Experimental): Participants in this group receive a single dose of TQ on Day 1 or Day 2 and a single dose of CQ daily, on Days 1 to 3.
  Interventions: Drug: Tafenoquine; Drug: Chloroquine
- PQ/CQ (Active Comparator): Participants in this group receive a single dose of PQ daily from Day 1 or 2, up to Day 14 (or Day 15 if PQ started on Day 2) and a single dose of CQ daily, on Days 1 to 3.
  Interventions: Drug: Primaquine; Drug: Chloroquine

INTERVENTIONS:
Drug: Tafenoquine — A single dose of TQ will be administered orally on Day 1 or Day 2.
  Arms: TQ/CQ
Drug: Primaquine — A single dose of PQ will be administered orally, daily, on Day 1 or 2 to Day 14 (or Day 15 if PQ started on Day 2).
  Arms: PQ/CQ
Drug: Chloroquine — A single dose of CQ will be administered orally, daily, on Days 1 to 3.

SUMMARY:
The aim of this study is to collect efficacy and safety data to support the registration of tafenoquine in India.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females >=2 years of age and under (<) 65 years of age, weighing >10 kg.
2. The participant has a positive malarial smear for P. vivax with a parasite density of >100/microliter and <100,000/microliter.
3. The participant has a screening Hb value >8 g/dL.
4. The participant has an axillary temperature of 37.5°C or history of fever 48 hours before recruitment.
5. The participant has a G6PD value (measured using the SD Biosensor STANDARDTM G6PD test) 6.1 units/gram (U/g) Hb for G6PD activity (6.1 U/g Hb cut-off is applicable for both males and females).
6. A female participant is eligible to participate if she is not pregnant or breastfeeding, and if one of the following conditions applies:

   * Is a woman of non-childbearing potential (WONCBP) as defined in
   * Is a Women of Childbearing Potential (WOCBP) and using a contraceptive method that is highly effective (with a failure rate of <1% per year), with low user dependency, during the study intervention period and for at least 90 days after the last dose of study intervention. The investigator should evaluate the potential for contraceptive method failure (e.g., noncompliance, recently initiated) in relationship to the first dose of study intervention. The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.
7. A WOCBP must test negative on a highly sensitive pregnancy test (urine or serum as required by local regulations) before the first dose of study intervention.
8. The participant is willing and able to comply with the procedures described in the study protocol. The participant or parent/legal guardian, as applicable, has given written informed, dated consent; and the participant has given written assent, if applicable, to participate in the study.

Exclusion Criteria:

1. The participant has severe P. vivax malaria as defined by WHO criteria [WHO, 2023].
2. The participant has a mixed malaria infection (identified by a malarial smear).
3. The participant has a condition that may affect absorption of study medication, such as severe vomiting (no food or inability to take food during the previous 8 hours).
4. The participant has a history of porphyria, psoriasis, or epilepsy.
5. The participant has a history of allergy, intolerance to or a known contraindication to the use of mefloquine (or other aryl amino alcohol drugs), chloroquine, tafenoquine, primaquine, any other 4- or 8-AQ or any of their respective excipients.
6. The participant has received treatment with any investigational drug within 30 days of study entry, or within 5 half-lives, whichever is longer.
7. The participant has previously enrolled in this study.
8. The participant has a recent history of illicit drug abuse or heavy alcohol intake that in the opinion of the investigator could compromise full participation in the study or adherence to study procedures.
9. Participants with a current or past history of serious psychiatric disorders.
10. The participant has a clinically significant concurrent illness (e.g., pneumonia, tuberculosis, meningitis, septicemia, dengue, coagulopathy, severe hemorrhage, or febrile convulsions prior to consent) or a pre-existing condition (e.g., renal disease, malignancy, or severe malnutrition according to WHO child growth standards) or systemic disease predisposing patients to suffer from granulocytopenia, such as rheumatoid arthritis and lupus erythematosus or severe ocular disease.
11. The participant is known to be HIV-infected and/or is currently on antiretroviral therapy.
12. The participant is regularly using drugs with hemolytic potential.
13. The participant has a QT corrected by Fridericia's formula (QTcF) >450 msec, evidence of bradycardia (<50 beats per min) or ventricular arrhythmias on the screening ECG, a history of cardiac disease (e.g., myocardial infarction, congenital heart disease, or arrhythmia), hypokalemia (<2.9 millimoles per liter [mmol/L]) or hyperkalemia (>=6.0 mmol/L) at Screening.
14. The participant has taken drugs with antimalarial activity (e.g., artemisinin-based combination therapies, mefloquine, primaquine, chloroquine, tafenoquine or any other 4-AQ) within 30 days prior to study entry.
15. The participant has taken or will likely require during the study the use of:

    1. Histamine-2 blockers (restricted to first 3 days whilst receiving CQ)
    2. Antacids (restricted to first 3 days whilst receiving CQ)
    3. Drugs of the biguanide class (i.e., phenformin, metformin, buformin)
    4. Anti-arrhythmic agents (i.e., dofetilide, procainamide, pilsicainide)
    5. Medications that prolong the QTc interval
16. The participant has liver transaminases (ALT/AST) >2 times the upper limit of normal (ULN).

Ages: 2 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-11-13 (Actual); Primary Completion 2026-05-25 (Estimated); Study Completion 2026-05-25 (Estimated)

PRIMARY OUTCOMES:
Number of participants remaining recurrence-free during the 6 months post-treatment and have a negative blood smear at the Month 6 (end of study [EOS]) visit | Up to Month 6
  Two consecutive negative blood smears between Day 2 and Day 8, no positive blood smear for P. vivax parasites at any point during the 6-month follow-up period, and a negative P. vivax smear at the 6-month assessment.

SECONDARY OUTCOMES:
Number of participants with clinically relevant hemolysis change from baseline | Up to Day 14
  A decrease in hemoglobin of greater than or equal to (>=) 30% or greater than (>) 3g/deciliter (dL) from baseline; or an overall drop in hemoglobin below 6.0 g/dL or complications thereof (e.g., required transfusions, acute renal failure) are considered clinically relevant hemolysis changes.
Time to recurrence of P. vivax malaria | Up to Month 6
  Recurrence is defined as a positive blood smear for P. vivax parasites within the 6-month follow-up period, after clearance of blood-stage parasitemia.
Number of participants with treatment emergent adverse events (TEAEs) up to Month 6 | Up to Month 6
  An adverse event (AE) is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Number of participants with TEAEs meeting >= Division of Acquired Immunodeficiency Syndrome (DAIDS) Grade 3 criteria | Up to Month 6
  Severity was graded according to DAIDS grading criteria, where Grade 1-mild, Grade 2-moderate, Grade 3-severe, Grade 4-potentially life-threatening, Grade 5-Death.
Number of participants with drug related TEAEs | Up to Month 6
  An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Number of participants with serious AEs (SAEs) | Up to Month 6
  A SAE is any untoward medical occurrence that results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization or result in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant.
Number of participants with AEs resulting in treatment discontinuation | Up to Month 6
  An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Number of participants with AEs leading to study withdrawal | Up to Month 6
  An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Number of participants with AEs considered to be hematologically related | Up to Month 6
  An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Number of deaths | Up to Month 6
Liver chemistry changes meeting Hy's criteria | Up to Month 6
  Hy's criteria cases were defined as any elevated alanine aminotransferase (ALT) >=3 times upper limit of normal (ULN) and total bilirubin >=2 times ULN or ALT >=3 times ULN and international normalized ratio (INR) >1.5.
Laboratory parameters meeting >= Division of AIDS (DAIDs) Grade 3 criteria | Up to Month 6
Vital sign parameters meeting >=DAIDs Grade 3 criteria | Up to Month 6
Number of participants with TEAEs up to Week 4 | Up to Week 4
  An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Change from baseline at each study visit for clinical chemistry parameters (ALT, AST, ALP) | At Days 5, 8, 15, 29, 60, 90, 120, 150 and 180
  Data for alanine aminotransferase (ALT), aspartate aminotransferase (AST) and alkaline phosphatase (ALP) is measured in international units/liter (IU/L).
Change from baseline at each study visit for clinical chemistry parameters (CPK) | At Days 5, 8, 15, 29, 60, 90, 120, 150 and 180
  Data for creatine phosphokinase (CPK) is measured in units per liter (U/L).
Change from baseline at each study visit for clinical chemistry parameters (total bilirubin, indirect bilirubin, blood urea nitrogen [BUN]/Urea, and serum creatinine) | At Days 5, 8, 15, 29, 60, 90, 120, 150 and 180
  Clinical chemistry parameters are measured in milligrams per decilitre (mg/dL).
Change from baseline at each study visit for clinical chemistry parameters (serum electrolytes) | At Days 5, 8, 15, 29, 60, 90, 120, 150 and 180
  Data for serum electrolytes is measured in millimoles per liter (mmol/L).
Change from baseline at each study visit for haematology parameters (platelet count) | At Days 5, 8, 15, 29, 60, 90, 120, 150 and 180
  Platelets are measured in number of platelets per microliter (µL).
Change from baseline at each study visit for haematology parameters (red blood cell [RBC] count) | At Days 5, 8, 15, 29, 60, 90, 120, 150 and 180
  Data for RBC is measured in millions of cells per microliter (number of RBCs x10^6/µL).
Change from baseline at each study visit for haematology parameters (mean corpuscular volume [MCV]) | At Days 5, 8, 15, 29, 60, 90, 120, 150 and 180
  Data for MVC is measured in femtoliters (fL).
Change from baseline at each study visit for haematology parameters (mean corpuscular hemoglobin [MCH]) | At Days 5, 8, 15, 29, 60, 90, 120, 150 and 180
  Data for MCH is measured in picograms (pg) per cell.
Change from baseline at each study visit for haematology parameters (percentage of reticulocytes) | At Days 5, 8, 15, 29, 60, 90, 120, 150 and 180
Change from baseline at each study visit for haematology parameters (white blood cell count [WBC] with differential) | At Days 5, 8, 15, 29, 60, 90, 120, 150 and 180
  Data for neutrophils, lymphocytes, monocytes, eosinophils and basophils is presented as a count, which measures a percentage (%) of the WBC.
Change from baseline at each study visit for haematology parameters (hemoglobin) | At Days 5, 8, 15, 29, 60, 90, 120, 150 and 180
  Hemoglobin is measured in grams per deciliter (g/dL).
Change from baseline at each study visit for haematology parameters (hematocrit) | At Days 5, 8, 15, 29, 60, 90, 120, 150 and 180
  Hematocrit is measured in volume percentage (%) of RBC in blood.

CONTACTS AND LOCATIONS:
Locations (4):
- India (4):
  - GSK Investigational Site, Ahmedabad
  - GSK Investigational Site, Kolkata
  - GSK Investigational Site, Mumbai
  - GSK Investigational Site, Surat

IPD SHARING:
Plan to Share IPD: Yes
GSK will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf